CLINICAL TRIAL: NCT01555021
Title: Pharmacogenomics for Antidepressant Guidance and Education
Status: Terminated | Type: Observational
Why Stopped: The study was an inpatient, but PI left inpatient at MGH on July 1, 2012
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John D. Matthews, Director of Research and Training, Massachusetts General Hospital
Other Study IDs: 2011-P-001921
Record Dates: First submitted 2012-02-16; First posted 2012-03-15 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-03

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Although the protocol included taking saliva samples from all subjects for GWAS analysis at a later date, GWAS analysis was not performed on any of the subjects due to the early termination of the study..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment as Usual (TAU): This group will provide blood samples to be analyzed at a later date for genotyping to determine the activity of CYP-450 enzymes that are important in metabolizing antidepressant medications.Treatment will be initiated based on the attending clinicians decision making absent genotyping results.
  All subjects in the group will receive the following assessment instruments for diagnosis: SCID-I/P and the Mini International Neuropsychiatric Interview (MINI)
  All subjects in the group will have the severity of their depression measured by the HAM D-17 (physician rating scale), the QIDS-SR-16 (patient rating). Clinical status will be measured by the CGI-S scale (1-7 with 7 being high functioning). Side effects ratings will be measured by the UKU. ATRQ will be used to assess the degree of treatment resistance by measuring the number of prior antidepressant trials.
  Patients in the TAU group will provide saliva samples for future GWAS analysis.
- Assay Guided Treatment (AGT): This group will provide blood samples for genotyping test to determine the activity of CYP-450 enzymes that are important in metabolizing antidepressant medications . This test result will be available within 3-5 days available to guide clinicians in their choice and dosing of antidepressant medications.
  All subjects in the group will have the severity of their depression measured by the Hamilton Depression Rating Scale-17 (physician rating scale), the QIDS-SR-16 (patient rating scale). Clinical status will be measured by the CGI-S scale (1-7 with 7 being high functioning). Side effects ratings will be measured by the Udvalg for Kliniske Undersogelser (UKU). ATRQ will be used to assess the degree of treatment resistance by measuring the number of prior antidepressant trials.
  Patients in the AGT group will provide saliva samples for future GWAS analysis.
  Interventions: Genetic: Genotyping assays

INTERVENTIONS:
Genetic: Genotyping assays — Patients will provide blood samples at the beginning of the study. If the patient is in the AGT group (as opposed to the TAU group), their blood samples will be sent for genotyping immediately. AGT psychiatrists will be given the results of genotyping within 3-5 days in order to decide which antidepressants to use long-term and at what doses. Patients in the Treatment as Usual group will have their blood samples stored for future analysis. Both groups will provide saliva samples for GWAS analysis at a alter date; however, since the study was terminated early, GWAS testing for both groups and genotyping for the TAU group were not performed.
  Patients will receive questionnaires to measure their mood, side effects, and symptoms.
  Patients will be asked to participate in 3 follow-up phone calls (1 month, 3 months, and 6 months) to measure their mood.
  Groups: Assay Guided Treatment (AGT)

SUMMARY:
More than one out of three individuals treated for major depressive disorder (MDD) do not experience a full reduction of symptoms even when treated with adequate antidepressant medication. These individuals may have treatment-resistant depression. This is a condition that contributes to the tremendous costs of MDD, in terms of health care costs, functional impairment (limitation of an individual's functional ability), and diminished quality of life.

There is a clear need for personalized medicine, for people at high risk for treatment-resistant depression. If these individuals could be identified early in the course of their depression, they could be recommended for more intensive or specialized interventions. Doing so could improve their likelihood of having a full reduction in their symptoms.

Today, there are many treatment options for MDD. Individuals can spend months or years in and out of treatment before receiving one that works for their treatment-resistant depression.

The investigators want to study treatment resistant depression by examining specific genes (genotyping) that might influence how your body responds to certain antidepressant medications. This process of examining specific genes is not experimental. To look at your specific genes, the investigators will collect a blood sample. Genes contain the material passed from parent to child that determines the make-up of the body and mind. For example, some genes control the color of your hair or eyes. Genes are contained in your DNA (deoxyribonucleic acid). There are many differences in DNA, from one person to another. These differences may affect a person's chances of having a particular disease.

DETAILED DESCRIPTION:
This will be a 6-month, randomized, controlled study of assay-guided treatment (AGT) versus treatment as usual (TAU) in adult inpatients with major depressive disorder. Two hundred subjects will be randomized to receive AGT or TAU. After subjects are screened, determined to be eligible, and complete baseline assessments, blood samples for genotyping will be obtained from all subjects as well as saliva samples for future GWAS analysis from all subjects. Only those subjects that are randomized to the AGT arm will have their blood samples immediately analyzed. Subjects in the TAU arm will have their blood samples stored for future analysis..

Once the blood samples are obtained, the attending psychiatrists will be asked to indicate their top three choices of antidepressants and at what doses they will initiate treatment. In order to prevent delays in providing treatments, the first choice antidepressants will be started prior to receiving assay results.

Upon receiving the assay reports (AGT arm), the attending psychiatrists will be asked whether the reports influenced their choice of antidepressant treatments and doses of antidepressants, as well as their confidence in their choices. The attending psychiatrists will then document any switches in antidepressant treatments or changes in doses of current antidepressant medications on a structured form. The assay reports will be available between 3 to 5 days after the blood samples are taken. The attending psychiatrists who are randomized to be provided the results of CYP genotyping will also be provided a phone number for consultation with Genomind Labs regarding the interpretation of the results.

Trough antidepressant blood samples for the AGT arm (10-12 hours after last dose) for therapeutic drug monitoring (TDM) will be obtained within 24 hours of discharge. Blood samples will also be obtained from the TAU arm, but they will be stored for future analysis of CYP genotyping and biomarker analysis of treatment resistant MDD. Clinical follow-up will proceed as felt to be clinically indicated. For subjects who have been discharged before the assay results are received, the attending psychiatrists will complete the from indicating changes in treatments as if patients were still in hospital. Results and recommendations will be forwarded to the identified outpatient psychiatrists. (note: blood levels of antidepressants were not analyzed)

The AGT arm is not standard care for patients with depression. The addition of assay-results and questionnaires makes the AGT arm different than standard care. Only the questionnaires make the TAU arm different than standard care.

Note:

Within 24 hours after you are admitted to the Inpatient Psychiatric Unit, the "baseline" assessment will occur. If you stay in the Inpatient Psychiatric Unit for more than one week, the "weekly" assessment will occur every 7 days. Typically, patients spend an average of 8-10 days in the Inpatient Psychiatric Unit. The day before or the day of your discharge from the Inpatient Psychiatric Unit, your "discharge" assessment will occur. One, 3, and 6 months after you are discharged, you will be asked to complete follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Written informed consent
* Meets DSM-IV criteria in the Structured Clinical Interview for DSM-IV-TR (SCID-I/P)17 and the MINI for current major depressive disorder, without psychotic features
* QIDS-SR score of at least 10 (i.e., moderate depression) at initial visit
* Failure of at least 1 prior adequate trial of a standard antidepressant (i.e., 6 weeks at adequate dose), assessed by the Antidepressant Treatment History Questionnaire (ATRQ)18 criteria
* Inpatient and expected to remain so for 5 or more days
* Hospitalized within past 72 hours

Exclusion Criteria:

* Pregnant women or women of child bearing potential who are not using a medically accepted means of contraception (to include oral contraceptive or implant, condom, diaphragm, spermicide, intrauterine device, tubal ligation, or partner with vasectomy). Immediately after the pregnancy test, women with positive pregnancy tests will be unable to enroll in the study
* Women who are breastfeeding
* Patients who have taken an investigational psychotropic drug within the last 3 months
* Section 12 status (involuntary admission)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was conducted on the 24-bed inpatient psychiatric unit at Massachusetts General Hospital. Written informed consent was obtained using the MGH-IRB approved consent form. A competency assessment consisting of four questions about the study was obtained. All subjects received a comprehensive psychiatric and medical evaluation including a comprehensive metabolic panel, TSH B12, folic acid, lipid panel and a urine pregnancy test for women of child-bearing age. Subjects needed to meet DSM-IV criteria for major depressive disorder.
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Matthews, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although clinicians were randomized to either receive or not receive the AGT results, they were not considered enrolled. Only the patients were enrolled in the study. Also, each participating clinician covered only one subject.
Groups:
- Treatment as Usual: Subjects will provide blood samples prior to treatment, but will have their blood stored for later analysis.
  Subjects will receive questionnaires to measure their mood, side effects, and symptoms.
  Subjects will provide a saliva samples for GWAS analyses at a later date. However, the GWAS analyses were not performed due to the early termination of the study.
- Assay Guided Treatment: This test is used to guide clinicians in their recommendation antidepressant drugs based on CYP 450 gene activity for 1A2, 2C9, 2C19, 2D6, and 3A/4.
  Subjects will be asked to provide blood samples. For subjects in the Assay-Guided Treatment group, their blood will be genotyped. Their psychiatrists will be given the results of the tests and then they will decide which antidepressants to use.
  Subjects will receive questionnaires to measure their mood, side effects, and symptoms.
  Subjects will be asked to provide saliva samples for GWAS analysis at a later date; however, GWAS analysis was not performed due to early termination of the study.
Period: Overall Study
Arm/Group | Treatment as Usual | Assay Guided Treatment
Started | 2 | 2
Completed | 1 (One treatment as usual subject completed 1 month, 3 month, and 6 month follow up visits) | 0 (None of the AGT subjects competed month 1, month 3, or month 6 follow up visits.)
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Treatment as Usual: Subjects in the Treatment as Usual group will proceed with treatment as usual, but have their blood samples for genotyping stored for future analysis.
  Patients will receive questionnaires to measure their mood, side effects, and symptoms.
  Subjects will be asked to provide saliva samples for GWAS analysis at a later date (note: GWAS analysis and genotyping for the Treatment as Usual group was not performed due to early termination of the study)
  Patients will be asked to participate in 3 follow-up phone calls to measure their mood.
- Assay Guided Treatment: This group will receive a genotyping test to determine the specific levels of gene activity. This test was used to guide clinicians decision making for which antidepressants to prescribe and/or at what doses.
  Subjects will receive questionnaires to measure their mood, side effects, and symptoms.
  Subjects will be asked to provide saliva samples for GWAS analysis at a later date (note; GWAS analysis was not performed in the AGT group due to early termination of the study.
  Subjects will be asked to participate in 3 follow-up phone calls to measure their mood.
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual | Assay Guided Treatment | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 59 [57 to 61] | 43.5 [25 to 62] | 51.25 [25 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Quick Inventory of Depressive Symptoms-Self Rating (SR) 16 Item
Description: To determine the efficacy of assay-guided treatment (AGT) versus treatment-as-usual (TAU), in terms of depression severity as measured by change in the Quick Inventory of Depressive Symptoms (QIDS-SR 16), adjusted for baseline severity, upon discharge, and at 1, 3, and 6 months post discharge from inpatient treatment. The QUIDS-SR 16 is a self rating 16 item multiple-choice questionnaire that measure severity of depression over the past week. The range on the QIDS-SR IS 0-27, with 0-5 indicating no depression; 6-10, mild depression; 11-15; moderate depression; 16-20 severe depression; and greater than or equal to 21, very severe depression.
Time Frame: Measured: Baseline (within 72 hours of admission), once weekly (+/- 24 hours), discharge (7-10 days after admission +/- 24 hours), and 1, 3, 6 months after discharge (+/- 4 weeks)
Population: Quick Inventory of Depression symptom-16 (QIDS-SR 16) Baseline. Data was not collected for all time points for all participants.
Measure: Mean (Full Range); unit: Score on QIDS-SR
Groups:
- Treatment as Usual: Subjects will be asked to provide blood samples for CYP 450 genotyping; however, the genotyping analysis will occur at a later date.
  Subjects will receive questionnaires to measure their mood, side effects, and symptoms.
  Subjects will be asked to provide a saliva sample for GWAS analysis at a later date. (note: genotyping analysis and GWAS analysis was not performed due to early termination of the study)
- Assay Guided Treatment: This test is used to guide clinicians in their recommendations for antidepressant drugs based on CYP 450 gene activity for 1A2, 2C9, 2C19, 2D6, and 3A/4.
  Subjects will be asked to provide a blood samples for CYP 450 genotyping. Subjects in the Assay-Guided Treatment group, will have their blood samples genotyped immediately. Their psychiatrists will be given the results of the tests within 3 to 5 days and then they will decide which antidepressants to use.
  Subjects will receive questionnaires to measure their mood, side effects, and symptoms.
  Subjects will be asked to provide a saliva sample for GWAS analysis at a later date. (note: GWAS analysis was not performed due to early termination of the study)
Arm/Group | Treatment as Usual | Assay Guided Treatment
Number analyzed (Participants) | 2 | 2
Score on QIDS-SR
  QIDS-SR 16 Baseline | 18 [17 to 19] | 22.5 [18 to 27]
  QIDS 16 Discharge: number analyzed (Participants) | 2 | 0
  QIDS 16 Discharge | 7.5 [6 to 9] |
  QIDS 16 at 1 month: number analyzed (Participants) | 1 | 0
  QIDS 16 at 1 month | 6 [6 to 6] |
  QIDS 16 at 3 months: number analyzed (Participants) | 1 | 0
  QIDS 16 at 3 months | 4 [4 to 4] |
  QIDS at 6 months: number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Clinician's Report That AGT Modified His/Her Decision Regarding Which Antidepressant to Prescribe.
Description: Clinicians randomized to receive AGT results were asked to report whether the AGT results impacted their decision making with regards to their choice of antidepressant and/or dosing of the antidepressant.
Time Frame: Measured: +/- 24 hours of baseline assessments and +/- 24 hours of receiving assay results
Population: 2 of 4 clinicians received AGT results for antidepressant decision making. One of two clinicians randomized to receive AGT results reported that his choice of antidepressant was definitely influenced by AGT results; the other clinician randomized to receive AGT results did not receive the AGT information within the defined time limit.
Measure: Number; unit: participants
Groups:
- Treatment as Usual: Subjects will provide a blood sample for CYP-450 genotyping; however, the Treatment as Usual group will have their blood samples stored for analysis at a later date..
  Patients will receive questionnaires to measure their mood, side effects, and symptoms.
  Subjects will provide a saliva sample for GWAS analysis at a later date. (note: genotyping and GWAS analysis were not performed on any subjects due to early termination of the study)
- Assay Guided Treatment: This test is used to guide clinicians in their recommendation antidepressant drugs based on CYP 450 gene activity for 1A2, 2C9, 2C19, 2D6, and 3A/4.
  Subjects will be asked for a blood sample for CYP-450 genotyping. If the patient is in the Assay-Guided Treatment group, their blood will be genotyped immediately. Their psychiatrists will be given the results of the tests within 3 to 5 days and then they will decide whether to change their original first choice antidepressants.
  Patients will receive questionnaires to measure their mood, side effects, and symptoms.
  Subjects will provide a saliva sample for GWAS analysis at a later date. (note: GWAS analysis was not performed on any subjects due to early termination of the study)
Arm/Group | Treatment as Usual | Assay Guided Treatment
Number analyzed (Participants) | 0 | 2
participants
  AGT beneficial in decision making: number analyzed (Participants) | 0 | 1
  AGT beneficial in decision making |  | 1
  AGT not beneficial in decision making: number analyzed (Participants) | 0 | 1
  AGT not beneficial in decision making |  | 0

3. Secondary Outcome: Treatment Adherence
Description: To determine the impact on adherence of AGT versus TAU at 7-10 days after admission
Time Frame: To determine the impact on adherence of AGT versus TAU at 7-10 days after admission
Population: Number of subjects adherent to antidepressant medications
Measure: Count of Participants; unit: Participants
Groups:
- Treatment as Usual: Subjects who are in the Treatment as Usual group will provide blood samples for genotyping, but their blood samples will be stored for analysis at a later date.
  Subjects will receive questionnaires to measure their mood, side effects, and symptoms.
  Subjects will provide a saliva sample for GWAS analysis at a later date. (note: genotyping for CYP 450 and GWAS analysis were not performed due to early termination of the study).
- Assay Guided Treatment (AGT): Subjects will provide a blood sample. Subjects in the AGT group will have their blood samples genotyped immediately. The treating psychiatrists will be given the results of the tests in 3 to 5 days and then they will decide whether to continue or change their first choice antidepressants. The genotyping test is a one-time occurrence that happens at the beginning of the study.
  Subjects will receive questionnaires to measure their mood, side effects, and symptoms.
  Subjects will provide a saliva sample for GWAS analyses at a later date. (note: GWAS analyses were not performed due to early termination of the study).
Arm/Group | Treatment as Usual | Assay Guided Treatment (AGT)
Number analyzed (Participants) | 2 | 2
Participants
  Number adherent at discharge | 2 | 2
  Number adherent at 1 month: number analyzed (Participants) | 1 | 0
  Number adherent at 1 month | 1 |
  Number adherent at 3 months: number analyzed (Participants) | 1 | 0
  Number adherent at 3 months | 1 |
  Number adherent at 6 months: number analyzed (Participants) | 1 | 0
  Number adherent at 6 months | 1 |

4. Secondary Outcome: Adverse Events (Side Effects)
Description: To determine the impact of AGT versus TAU on total number of side effects determined by using the Udvalg for Kliniske Undersogelser (UKU).
  1. TAU group reported a total of 8 different side effects, but 11 total events with two subjects over the time frame listed below; the events were expected. (see itemized adverse events)
  2. AGT group reported a total of four different side effects and 4 events with one subject over the time frame listed; the events were expected.(see itemized adverse events)
Time Frame: Measures at discharge, 1 month, 3 months, and 6 months
Population: Missing data on one AGT subjects
Measure: Number; unit: Number of side effects
Groups:
- Treatment as Usual: This test is used to guide clinicians in their recommendation antidepressant drugs based on CYP 450 gene activity for 1A2, 2C9, 2C19, 2D6, and 3A/4.
  Subjects in this group will be asked to provide blood samples for CYP genotyping at a later date. Their psychiatrists will decide which antidepressants to use as usual.
  Subjects will receive questionnaires to measure their mood, side effects, and symptoms.
  Subjects will be asked to provide saliva samples for GWAS analysis at a later date. (note: CYP genotyping and GWAS analysis for this group was not performed due to early termination of the study).
- Assay Guided Treatment: This test is used to guide clinicians in their recommendation antidepressant drugs based on CYP 450 gene activity for 1A2, 2C9, 2C19, 2D6, and 3A/4.
  Subjects will be asked to provide blood samples for CYP 450 genotyping.Their psychiatrists will be given the results of the tests within 3 to 5 days and then they will decide which antidepressants to use.
  Subjects will receive questionnaires to measure their mood, side effects, and symptoms.
  Subjects will provide a saliva sample for GWAS analysis at a later date. (note: GWAS analysis was not performed on any subjects due to early termination of the study).
Arm/Group | Treatment as Usual | Assay Guided Treatment
Number analyzed (Participants) | 2 | 1
Number of side effects
  Number of side effects at discharge | 7 | 4
  Number of side effects at 1 month: number analyzed (Participants) | 1 | 0
  Number of side effects at 1 month | 1 |
  Number of side effects at 3 months: number analyzed (Participants) | 1 | 0
  Number of side effects at 3 months | 1 |
  Number of side effects at 6 months: number analyzed (Participants) | 1 | 0
  Number of side effects at 6 months | 2 |

ADVERSE EVENTS:
Time Frame: Six months for one subject in the TAU group. Up to 2 weeks for two AGT subjects and one TAU subject. These subjects did not complete 1 month, 3 month, or 6 month follow up visits due to lost to follow up and early termination of the study.
Description: There were no all cause mortality or serious adverse events. All adverse events were expected and measured using the Udvalg for Kliniske Undersogelser (UKU).
Groups:
- Treatment as Usual (TAU): Patients in the TAU group provided blood samples to obtain genotyping to determine the specific activity of genes important in metabolizing antidepressants and to be processed at a later date; however, these blood samples were not analyzed due to the early termination of the study.
  Patients received questionnaires to measure their mood, side effects, and symptoms.
  Patients provided a saliva sample for GWAS analysis at a later date; however, GWAS analysis was not done due to the early termination of the study.
- Assay Guided Treatment (AGT): Patients in the AGT provided blood samples to obtain genotyping to determine the specific activities of genes important in metabolizing antidepressants. This test was used, at the beginning of treatment to guide clinicians in making recommendations as to which antidepressants and at what doses to prescribe.
  Patients received questionnaires to measure their mood, side effects, and symptoms.
  Patients in the AGT group provided saliva samples for GWAS analysis; however, GWAS analysis was not done due to the early termination of the study.
Arm/Group | Treatment as Usual (TAU) | Assay Guided Treatment (AGT)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment as Usual (TAU) (N=2) | Assay Guided Treatment (AGT) (N=2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 1 (1) | 1 (1)
Reduced sexual desire (General disorders) | 1 (1) | 1 (1)
Increased dreaming (Psychiatric disorders) | 1 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
weight gain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Increased appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased sleep (Psychiatric disorders) | 1 (1) | 1 (1)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No